CLINICAL TRIAL: NCT03994276
Title: The Postprandial Effects After Consumption of Chick-Pea Oral Doses on Glucose, Insulin, and Gut Hormone Responses. The PEA-POD Study
Brief Title: The Postprandial Effects of Chick-Pea Consumption on Glucose, Insulin, and Gut Hormone Responses (PEA-POD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Quadram Institute Bioscience (Other); New-Food Innovation (Unknown); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HR-18/19-8431
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-06

CONDITIONS: Postprandial Period
Keywords: Chickpea; Cell Wall; Dietary Fibre; Postprandial; Metabolism; Enteroendocrine

STUDY DESIGN:
Intervention Model Description: Cross-over design: Each participant will receive a control plus 2 treatments
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase 1: Control (Placebo Comparator): oral glucose tolerance test (OGTT): 58g Dextrose in 330ml water
  Interventions: Dietary Supplement: Chickpea powder
- Phase1: Chickpea Control (Active Comparator): "sub-cellular" Chickpea powder: 58g total available carbohydrate, provided as 50g from chickpea powder + 8g from chocolate flavouring
  Interventions: Dietary Supplement: Chickpea powder
- Phase1: Chickpea Powder (Experimental): Chickpea powder: 58g total available carbohydrate, provided as 50g from chickpea powder + 8g from chocolate flavouring
  Interventions: Dietary Supplement: Chickpea powder
- Phase 2: Control (Active Comparator): Wheat bread: breakfast consisting of a 100% wheat bread roll containing 54g available carbohydrate + 20g diabetic strawberry jam containing 2g sugar + 360ml water
  Interventions: Dietary Supplement: Chickpea powder
- Phase 2: 30%Chickpea Powder (Experimental): Wheat bread: breakfast consisting of a 70% wheat / 30% Chickpea powder bread roll containing 54g available carbohydrate + 20g diabetic strawberry jam containing 2g sugar + 360ml water
  Interventions: Dietary Supplement: Chickpea powder
- Phase 2: 60%Chickpea Powder (Experimental): Wheat bread: breakfast consisting of a 40% wheat / 60% Chickpea powder bread roll containing 54g available carbohydrate + 20g diabetic strawberry jam containing 2g sugar + 360ml water
  Interventions: Dietary Supplement: Chickpea powder

INTERVENTIONS:
Dietary Supplement: Chickpea powder — Chickpea powder is produce using novel production techniques to maintain chickpea cell structure. It will be incorporated into a drink (Dextrose control), or baked into bread rolls at 30% or 60% substitution of wheat flour(100% Wheat flour control).

SUMMARY:
Pulses have a high fibre content, contribute to lowering fasting blood cholesterol levels and improving glycaemic control, and have shown also considerable promise in supporting the dietary management of cardiovascular disease (CVD), type-2 diabetes mellitus (T2DM) and obesity. It is now established that cellular integrity (maintenance of cell wall structure) is a key factor responsible for the low glycaemic index (GI) of pulses. The maintenance of the cell wall structure restricts starch digestion and therefore glucose production in the gut. Thus, cell damage results in a loss of such properties and also the potential health benefits to consumers.

This knowledge has presented an opportunity to exploit alternative processing techniques for the manufacture of pulse-based ingredients. We have successfully created a dry powder consisting predominantly of intact cells which still retains low digestibility (>60% resistant starch). This chickpea powder (CPP) was found to be stable under long-term storage, has a neutral taste and aroma, and showed promise as a low GI 'flour-substitute'.

This study will investigate blood sugar, insulin and gut hormone levels (post-prandial glycaemic, insulinaemic and hormone responses) following the consumption of CPP consumed at breakfast, as a drink and incorporated into a food matrix (bread).

DETAILED DESCRIPTION:
The nutritional and potential long-term health benefits of consuming pulses have been well documented. Pulses have a high fibre content, contribute to lowering fasting blood cholesterol levels and improving glycaemic control, and have shown also considerable promise in supporting the dietary management of cardiovascular disease (CVD), type-2 diabetes mellitus (T2DM) and obesity. They are gluten-free and are also an affordable and accessible source of starch, protein, and dietary fibre. It is now established that cellular integrity (maintenance of cell wall structure) is a key factor responsible for the low glycaemic index (GI) of pulses. The maintenance of the cell wall structure restricts starch digestion and therefore glucose production in the gut. Thus, cell damage (i.e. as occurs extensively during milling of pulses into flour) results in a loss of such properties and also the potential health benefits to consumers.

This knowledge has presented an opportunity to exploit alternative processing techniques for the manufacture of pulse-based ingredients that preserve the desirable low GI of whole pulses. Incorporation of such ingredients has the potential to lower the glycaemic and insulinaemic responses to staple food products and/or may promote satiety, thereby ameliorating the dietary management of T2D and obesity and reducing the risk factors associated with these diseases. Building on new understanding of the conditions required to preserve cellular integrity, we have successfully created a dry powder consisting predominantly of intact cells which still retains low digestibility (>60% resistant starch). This chickpea powder (CPP) was found to be stable under long-term storage, has a neutral taste and aroma, and showed promise as a low GI 'flour-substitute'.

This study will investigate blood sugar, insulin and gut hormone levels (post-prandial glycaemic, insulinaemic and hormone responses) following the consumption of CPP consumed as a drink and incorporated into a food matrix (bread). It is hypothesised that the structure of the CCP will result in a reduced post-prandial glycaemic response, while maintaining (or improving) the insulinaemic and gut hormone responses. This regulation of blood sugar levels following a meal would be beneficial for people with impaired glucose metabolism, such as T2DM. This study will consist of two phases, both utilising a three-arm, random crossover design.

Phase 1 aims to test the glucose response to unmodified CPP (i.e. has not been cooked). This will involve the consumption of the following test drinks containing 50g of available carbohydrate (i.e. starch and/or sugars): (1) Glucose (an oral glucose tolerance test, OGTT); (2) Control chickpea product (no cellular integrity); and (3) the CPP. These test drinks will be consumed in random order on three separate visits. In order to ensure the test carbohydrates remains in solution, all test drinks will be made up in an equivalent volume of 330 ml (bottled water) containing chocolate flavouring. Participants will be required to fast overnight, a capillary blood glucose measurement will be taken at t=0, followed by consumption of the test drink within 5 min. Further capillary blood glucose measurements will be taken at t=10, 20, 30, 45, 60, 90, and 120 min. Additionally, participants will be provided with a Constant Glucose Monitor (CGM) that will be applied to the upper arm 24hrs prior to the first study day. All three study visits will be completed in 12 days (The length of CGM activity). It is hypothesised that the cell wall integrity in the CPP drink will result in a reduced post-prandial glycaemic response compared to the control chickpea product and the OGTT standard.

Outcome measures: The primary outcome of Phase 1 will be the glycaemic response to the consumption of CPP drink compared to both the OGTT and control chickpea product. In vitro studies suggest that maintenance of cellular integrity will reduce the early phase of post-prandial glycaemia, as assessed by the incremental area under the curve (iAUC) iAUC0-60min and maximum blood glucose concentration (Cmax). Secondary measures such as the time to reach maximum blood glucose concentration (Tmax), iAUC0-120min and iAUC60-120min will also be assessed.

Phase 2 aims to test the glucose, insulin and gut hormone response to CPP incorporated into a staple food. This will involve the consumption of wheat-based breads containing 50g of available carbohydrate and either; (1) wheat bread (control) (2) wheat bread with 30% CPP substitution of wheat flour, and (3) wheat bread with 60% CPP substitution of wheat flour. These breads will be consumed as part of a breakfast following an overnight fast on three separate study visits. Post-prandial concentrations of plasma glucose, insulin, glucose-dependent insulinotropic peptide (GIP), glucagon-like peptide 1 (GLP-1), peptide YY (PYY) and C-peptide will be measured; at commencement of meal, t=0, and following consumption at, t=15, 30, 45, 60, 90, 120, 180, and 240 min. Additionally, participants will be provided with a Constant Glucose Monitor (CGM) that will be applied to the upper arm 24hrs prior to each study day.

Outcome measures: The primary outcome of Phase 2 will be iAUC0-60min for plasma glucose concentrations and corresponding plasma insulin/C-peptide responses, demonstrating the ability of cell wall integrity to limit starch digestion, and therefore, the rate of glucose appearance in the blood in the early phase of post-prandial glycaemia. Secondary outcome variables include iAUC0-120min, iAUC0-240min, 30-90 and 90-240, Cmax, Tmax changes from baseline up to 240 min for plasma glucose, insulin, and C-peptide concentrations. For the gut hormones plasma GIP, PYY and GLP-1 concentrations will be assessed using the same outcome variables. Subjective measures of study meals and ad libitum meal palatability will be collected at t=10 min and post lunch, respectively. Subjective measures of mood, satiety and digestive comfort will be collected t=0, 10, 30, 60, 120, 180, 210, 240 min and post lunch. The energy intake from the ad libitum lunch provided following the experimental period will also be compared. Subjective measures will be summarised using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 y
* Men and women
* Healthy (free of diagnosed diseases listed in the exclusion criteria)
* Body Mass Index 18-35 kg/m2
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed written consent

Exclusion Criteria:

* Those with known or suspected food allergies (particularly to wheat, as specified in the screening questionnaire and participant information form) or hypersensitivity
* Women who are pregnant, intending to become pregnant, or breastfeeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months.
* Body mass index <18 or >35 kg/m2
* Full Blood Counts and Liver Function test results outside of the normal range.
* Current smokers, or reported giving up smoking within the last 6 months History of substance abuse or alcoholism
* Reported history of Cardiovascular disease, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function)
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.8 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study: alpha-glucosidase inhibitors (acarbose:

Glucobay), insulin- sensitising drugs (metformin: Glucophage, Glucophage SR, Eucreas, Janumet; thiazolidinediones: Actos, Competact), sulfonylureas (Daonil, Diamicron, Diamicron MR, Glibenese, Minodiab, Amaryl Tolbutamide), and lipid- lowering drugs (statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates).

Other medications should be reviewed by a medical representative from KCL on a case by case basis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Phase 1: Postprandial Glycaemia (iAUC 0-60min) | 60 min
  The primary endpoint is iAUC 0-60 min for plasma glucose concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (iAUC 0-60min) | 60 min
  The primary endpoint is iAUC 0-60 min for plasma glucose, Insulin, c-peptide and Gut hormone concentrations

SECONDARY OUTCOMES:
Phase 1: Postprandial Glycaemia (iAUC 0-120min) | 120 min
  iAUC 0-120 min for plasma glucose concentrations
Phase 1: Postprandial Glycaemia (iAUC 60-120min) | 60 min
  iAUC 60-120 min for plasma glucose concentrations
Phase 1: Postprandial Glycaemia (Cmax) | 120 min
  Cmax for plasma glucose concentrations
Phase 1: Postprandial Glycaemia (Tmax) | 120 min
  Tmax for plasma glucose concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (iAUC 0-120min) | 120 min
  iAUC 0-120 min for plasma glucose, Insulin, c-peptide and Gut hormone concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (iAUC 0-240min) | 240 min
  iAUC 0-240 min for plasma glucose, Insulin, c-peptide and Gut hormone concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (iAUC 30-90min) | 60 min
  iAUC 30-90 min for plasma glucose, Insulin, c-peptide and Gut hormone concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (iAUC 90-240min) | 150 min
  iAUC 90-240 min for plasma glucose, Insulin, c-peptide and Gut hormone concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (Cmax) | 240 min
  Cmax for plasma glucose, Insulin, c-peptide and Gut hormone concentrations
Phase 2: Postprandial Glycaemia / Insulinaemia (Tmax) | 240 min
  Tmax for plasma glucose, Insulin, c-peptide and Gut hormone concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ellis, PhD, Principal Investigator — King's College London
Locations (1):
- Metabolic Research Unit, London, Please Choose, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bajka BH, Pinto AM, Perez-Moral N, Saha S, Ryden P, Ahn-Jarvis J, van der Schoot A, Bland C, Berry SE, Ellis PR, Edwards CH. Enhanced secretion of satiety-promoting gut hormones in healthy humans after consumption of white bread enriched with cellular chickpea flour: A randomized crossover study. Am J Clin Nutr. 2023 Mar;117(3):477-489. doi: 10.1016/j.ajcnut.2022.12.008. Epub 2022 Dec 28. PMID 36811474